CLINICAL TRIAL: NCT04571580
Title: Effect of Low-dose Intracoronary Reteplase During Primary Percutaneous Coronary Intervention on Myocardial Infarct Size in Patients With Acute Myocardial Infarction
Brief Title: Effect of Low-dose Intracoronary Reteplase on Myocardial Infarct Size During Primary Percutaneous Coronary Intervention
Acronym: RECOVERII
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study enrollment is slow due to the pandemic.
Sponsor: Ge Junbo (Other)
Responsible Party: Sponsor-Investigator, Ge Junbo, Director, Dept. of Cardiology, Zhongshan Hospital, Fudan University, Shanghai, China, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECOVERII
Record Dates: First submitted 2020-09-19; First posted 2020-10-01 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Acute ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Saline Solution; reteplase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): intracoronary infusion with saline
  Interventions: Drug: Normal Saline
- reteplase 9mg (Experimental): intracoronary infusion with reteplase 9mg
  Interventions: Drug: Reteplase Injection 9mg
- reteplase 18mg (Experimental): intracoronary infusion with reteplase 18mg
  Interventions: Drug: Reteplase Injection 18mg

INTERVENTIONS:
Drug: Normal Saline — intracoronary infusion with normal saline
  Other Names: intracoronary normal saline
  Arms: placebo
Drug: Reteplase Injection 9mg — low-dose intracoronary fibrinolytic therapy with reteplase 9mg
  Other Names: intracoronary reteplase 9mg
  Arms: reteplase 9mg
Drug: Reteplase Injection 18mg — low-dose intracoronary fibrinolytic therapy with reteplase 18mg
  Other Names: intracoronary reteplase 18mg
  Arms: reteplase 18mg

SUMMARY:
OBJECTIVE: To determine whether a therapeutic strategy involving low-dose intracoronary fibrinolytic therapy with reteplase infused after coronary reperfusion will reduce the myocardial infarction size.

DESIGN, SETTING, AND PARTICIPANTS: 306 patients presenting at 15 hospitals in China within 12 hours of acute ST-segment elevation myocardial infarction (STEMI) due to a proximal-mid-vessel occlusion of left anterior descending (LAD) coronary artery occlusion will be randomized in a 1:1:1 dose-ranging trial design. Patients will be followed up to 1 month.

INTERVENTIONS: Participants will be randomly assigned to treatment with placebo (n = 102), reteplase 9mg (n = 102), or reteplase 18mg (n = 102) by manual infusion over 2 minutes after reperfusion of the infarct-related coronary artery and before stent implant.

MAIN OUTCOMES AND MEASURES The primary outcomewas the myocardial infarct size (% left ventricular mass) demonstrated by contrast-enhanced cardiac magnetic resonance imaging (MRI) conducted from days 2 through 7 after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Acute STEMI with persistent ST-segment elevation or recent left bundle-branch block with a symptom onset to reperfusion time of 12 hours or less.
2. Angiographic criteria included a proximal-mid coronary artery occlusion (TIMI coronary flow grade 0 or 1) or, impaired coronary flow (TIMI flow grade 2, slow but complete filling) in the presence of definite angiographic evidence of large thrombus (TIMI grade ≥2) in left anterior descending (LAD) coronary artery.

Exclusion Criteria:

1. Rescue PCI after thrombolytic therapy.
2. Need for emergency coronary artery bypass grafting.
3. Presence of cardiogenic shock.
4. Life expectancy of < 6 months.
5. Inability to provide informed consent.
6. Contraindications for the use of thrombolysis, including active internal bleeding, history of intracranial haemorrhage or ischaemic stroke within 6 months, recent major surgery or trauma, severe uncontrolled hypertension, thrombocytopenia and severe liver or kidney failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size | from days 2 through 7 after enrollment
  Myocardial infarct size (% left ventricular mass) demonstrated by contrast-enhanced cardiac magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Amount of microvascular obstruction | from days 2 through 7 after enrollment
  The amount of microvascular obstruction (% of left ventricular mass) demonstrated by late gadolinium-enhanced MRI
ST-segment resolution | 60 minutes after reperfusion
  The percentage ST-segment resolution on an electrocardiogram
CKMB level | immediately before reperfusion (0 hours) and then again at 2 hours and at 24 hours
  CKMB area under the curve (AUC)
Left ventricular ejection fraction | 1 and 30 days after PCI
  Left ventricular ejection fraction assessed by echocardiography
Incidence of major adverse cardiac events (MACE) | 30 days after PCI
  The composite of cardiac mortality, nonfatal myocardial reinfarction and target vessel revascularization
Myocardial Blush Grade | 0-1 hour at the end of PCI
  Angiographic measures of reperfusion. The score goes from 0 to 3, with 3 being normal and 0 being absence of myocardial blush
TIMI corrected frame count | 0-1 hour at the end of PCI
  Angiographic measures of reperfusion. Thrombolysis in myocardial infarction score with corrected frame count from angiogram to assess myocardial perfusion
TIMI flow grade | 0-1 hour at the end of PCI
  Angiographic measures of reperfusion. The score goes from 0 to 3, with 3 being normal and 0 being absence of coronary flow

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Principal Investigator — Department of Cardiology, Zhongshan Hospital
Locations (1):
- Department of Cardiology, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Huang D, Ma Y, Wu H, Zhong X, Gao W, Zhou J, Qian J, Ge J. Impact of intracoronary reteplase during primary percutaneous coronary intervention on infarct size in large anterior myocardial infarction: rationale and design of the RECOVER II trial. Cardiovasc Diagn Ther. 2022 Jun;12(3):352-359. doi: 10.21037/cdt-21-756. PMID 35800360